CLINICAL TRIAL: NCT01966393
Title: An Open-label, Randomized, Three-way, Cross-over Study to Assess the Efficacy of Single-hormone Closed-loop Strategy, Dual-hormone Closed-loop Strategy and Conventional Insulin Pump Therapy in Regulating Glucose Levels During 60 Hours in Free-living Conditions in Patients With Type 1 Diabetes
Brief Title: Closed-loop Control of Glucose Levels (Artificial Pancreas) for 60 Hours in Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate Professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-07
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Hypoglycemia; Insulin; Glucagon; Closed-loop strategy; Artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dual-hormone closed-loop strategy (Active Comparator): In dual-hormone closed-loop strategy, variable subcutaneous insulin and glucagon infusion rates will be used to regulate glucose levels
  Interventions: Other: 60-hours intervention
- Single-hormone closed-loop strategy (Active Comparator): In single-hormone closed-loop strategy, variable subcutaneous insulin infusion rate will be used to regulate glucose levels
  Interventions: Other: 60-hours intervention
- Conventional insulin pump therapy (Active Comparator): In control visit, subjects will use conventional pump therapy to regulate glucose levels.
  Interventions: Other: 60-hours intervention

INTERVENTIONS:
Other: 60-hours intervention — Interventions will be conducted at the research centre (RC) or at the patient's home based on the patient's preference. If the study takes place at the RC, patients will be admitted at 7:00. If the study takes place at the patient's home, a research team member will be at the patient's home at 7:00. Closed-loop strategy will start at 8:00 on day 1 and end at 20:00 on day 3. During the interventions conducted at the RC, patients will have access to entertainment activities such as movies, video games, board games, foosball, etc. During the interventions conducted at the patient's home, patients will do their usual activities. For interventions conducted at the RC, patients will freely choose their meals from a large choice of prepared frozen meals. For interventions conducted at the patient's home, patients will freely choose their meals. Participants will be encouraged to conduct their usual physical activities whether they conduct the study at the RC or at the patient's home.

SUMMARY:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings. A dual-hormone closed-loop strategy would regulate glucose levels through the infusion of two hormones: insulin and glucagon.

The main objective of this project is to compare the efficacy of single-hormone closed-loop strategy, dual-hormone closed-loop strategy and conventional insulin pump therapy to regulate glucose levels in a 60-hours in non-standardized conditions in adults with type 1 diabetes.

The investigators hypothesized that 1) Controlling glucose levels using single- or dual-hormone CLS is feasible in free-living conditions for long period of time (60 hours); 2) Dual-hormone CLS is superior to single-hormone CLS as assessed by reducing time spent in hypoglycemic range; 3) Both single-hormone and dual-hormone CLS are superior to conventional pump therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of old.
* Clinical diagnosis of type 1 diabetes for at least one year.
* The subject will have been on insulin pump therapy for at least 3 months.
* HbA1c ≤ 12%.

Exclusion Criteria:

* Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
* Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
* History of pheochromocytoma or insulinoma (glucagon could induce an hormonal response of these tumors)
* Beta-blockers at high dose based on investigator's evaluation of dosage interference with glucagon (glucagon can modify effect of beta-blockers, mostly evident at very high doses)
* Chronic indometacin treatment (can prevent glucagon effect on liver thus its ability to raise glucose)
* Warfarin chronic treatment if INR monitoring cannot be evaluated (can increase the risk of bleeding)
* Anticholinergic drug (risk of interaction)
* Pregnancy.
* Severe hypoglycemic episode within two weeks of screening.
* Current use of glucocorticoid medication (except low stable dose and inhaled steroids).
* Known or suspected allergy to the trial products or meal contents (gluten free menus will be available).
* Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator (e.g. need for major revision of carbohydrate counting).
* Anticipating a significant change in exercise regimen between admissions (i.e. starting or stopping an organized sport).
* Failure to comply with team's recommendations (e.g. not willing to eat meals/snacks, not willing to change pump parameters, etc).
* Treatments that could interfere with glucagon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percentage of time of glucose levels (as measured by continuous glucose sensor) spent in the hypoglycemic range. | 60 hours
  Hypoglycemic range is defined to be between below 4 mmol/L

SECONDARY OUTCOMES:
Percentage of time of glucose levels (as measured by continuous glucose sensor) spent in target range. | 60 hours
  Target range is defined to be between 4 and 10 mmol/L from 7:00 to 22:00 and between 4 and 8 mmol/L from 22:00 to 7:00.
Percentage of time of glucose levels spent below 3.5 mmol/L | 60 hours
Percentage of time of glucose levels spent below 3.3 mmol/L | 60 hours
Area under the curve of glucose values below 4.0 mmol/L | 60 hours
Area under the curve of glucose values below 3.5 mmol/L | 60 hours
Area under the curve of glucose values below 3.3 mmol/L | 60 hours
Percentage of time of glucose levels spent above 8.0 mmol/L | 60 hours
Percentage of time of glucose levels spent above 10.0 mmol/L | 60 hours
Mean value of glucose levels | 60 hours
Standard deviation of glucose levels | 60 hours
Total insulin delivery | 60 hours
Number of patients with at least one hypoglycemic event with or without symptoms below 3.0 mmol/L based on glucose sensor reading | 60 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD, PhD, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada